CLINICAL TRIAL: NCT00012961
Title: Improving Health Services for Veterans With Schizophrenia
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Maryland, Baltimore County (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: VCR 99-012
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
Schizophrenia exacts a high toll on the lives of patients and their families and constitutes a major health care cost. VISN 5 has placed special emphasis on improving care for veterans with severe mental disorders, an effort recently recognized by the VA as a Program of Excellence in the Care of Seriously Mentally Ill Veterans.

DETAILED DESCRIPTION:
Background:

Schizophrenia exacts a high toll on the lives of patients and their families and constitutes a major health care cost. VISN 5 has placed special emphasis on improving care for veterans with severe mental disorders, an effort recently recognized by the VA as a Program of Excellence in the Care of Seriously Mentally Ill Veterans.

Objectives:

This study is implementing a set of promising QOC methods for assessing QOC for schizophrenia in routine settings, using the evidence-based treatment recommendations developed under the AHCPR/NIMH-sponsored Schizophrenia Patient Outcomes Research Team (PORT).

Methods:

A random sample of 350 persons with a schizophrenia spectrum disorder is being drawn from the VISN 5 sites. Patients must have more than one outpatient contact during the preceding six months. Each subject will participate in two one-hour interviews, one at baseline and another six months later. An informant, psychiatrist, therapist, etc. will also be interviewed to help validate participant response.

Status:

Project work is ongoing.

ELIGIBILITY:
Inclusion Criteria:

Patients must be adults currently in treatment for an Axis I schizophrenia spectrum disorder (DSM295) at VA.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan S. Bellack, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States